CLINICAL TRIAL: NCT07163858
Title: Comparison of Hemodynamic Management by Postural Mobilization Versus Chemical Vasoconstriction Using Noradrenaline Exclusively in Off-pump Coronary Artery Bypass Graft Surgery: A Prospective, Randomized, Comparative, Single-center Study.
Brief Title: Postural Mobilization Compared to Noradrenaline Only in Off-Pump CABG Surgery
Acronym: OPTICAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Infirmerie Protestante de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPL/01-2024; ID-RCB: 2024-A00683-44 (Other: ANSM)
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease With Need for Bypass Surgery; Coronary Artery Disease(CAD); Coronary Artery Bypass; Off Pump Coronary Artery Bypass Graft; Off Pump Coronary Artery Bypass Surgery; Hemodynamic Management; Hemodynamic Optimization; Noradrenaline
Keywords: open-heart coronary bypass; passive leg raising; hemodynamic management; off-pump CABG surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single-site, prospective, interventional, single-blind randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural Group: hemodynamic management using postural mobilization (+/- noradrenaline) (Experimental): In order to manage hemodynamics, postural mobilization will be applied by raising legs passively up to a 45° angle prior to any drug use (noradrenaline). If passive leg raising is not sufficient, noradrenaline will be used to stabilize hemodynamics,.
  Interventions: Procedure: passive leg raising for hemodynamic management during open-heart coronary bypass grafting
- Control group: use of noradrenaline only (no postural mobilization) (Active Comparator): Noradrenaline will be used to manage hemodynamics. Passive leg raising will not be used in this group
  Interventions: Procedure: Use of Noradrenaline only in control group

INTERVENTIONS:
Procedure: passive leg raising for hemodynamic management during open-heart coronary bypass grafting — Passive leg raising will be used in the experimental group in order to manage hemodynamics: legs will be raised to an angle of approx. 45°
  Arms: Postural Group: hemodynamic management using postural mobilization (+/- noradrenaline)
Procedure: Use of Noradrenaline only in control group — Noradrenaline will be used for hemodynamic management. Passive leg raising will not be used in this group
  Arms: Control group: use of noradrenaline only (no postural mobilization)

SUMMARY:
This interventional prospective randomized study is designed to compare hemodynamic management using postural mobilization (+/- noradrenaline) versus noradrenaline only in patients undergoing open-heart coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
OPTICAB is a single-site study in France that aims to compare two hemodynamic management techniques during off-pump coronary artery bypass graft (CABG) surgery: postural mobilization (+/- noradrenaline) versus noradrenaline only. Primary objective is to evaluate how often noradrenaline is needed when managing hemodynamics using postural mobilization (passive leg raising) during off-pump CABG surgery. The study will also compare revascularization rate and post-operative complications among both groups, and assess perioperative hemodynamic management during the 30-day follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* patient requiring isolated coronary bypass surgery
* Elective procedure or medical emergency
* First cardiac surgery
* Patient with an EF ≥30%
* Mandatory affiliation to a social security system
* Signed informed consent form
* Suspension of renin-angiotensin system inhibitors and angiontensn-neprilysin receptor blockers and sartans the day before surgical procedure

Exclusion Criteria:

* Contraindication to an inotropic substance (only NA will be used)
* Contraindication to passive leg raising
* Patient in a life-threatening emergency
* History of cardiac surgery
* Bilateral iliac or common femoral artery occlusion
* EF < 30%
* Pregnancy and breastfeeding
* Renal failure (GFR < 40 ml/min/1.73 m²)
* Patient with bilateral thigh amputation
* Class III obesity BMI > 40 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Assess use of noradrenaline in the experimental group (postural mobilization) vs control group (NA only) for hemodynamic management during open-heart coronary bypass graft surgery. | From beginning to end of urgery

CONTACTS AND LOCATIONS:
Locations (1):
- Infirmerie Protestante de Lyon, Caluire-et-Cuire, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
A plan has not yet been decided